CLINICAL TRIAL: NCT05493631
Title: A Phase 1b, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous MG1113 in Patients With Severe Hemophilia
Brief Title: A Phase 1b Study to Assess the Safety, Tolerability, PK and PD of MG1113 in Hemophilia Patient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MG1113_HP_P0101
Record Dates: First submitted 2022-07-21; First posted 2022-08-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hemophilia
Keywords: MG1113; Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (2.0 mg/kg, once weekly) (Active Comparator): * Anti-tissue factor pathway inhibitor (TFPI) recombinant antibody
  * Each vial contains 1mL of study drug
  * The subjects will be treated with 2.0 mg/kg once weekly in cohort 1.
  Interventions: Biological: MG1113
- Cohort 2 (A mg/kg, once weekly) (Active Comparator): * Anti-tissue factor pathway inhibitor (TFPI) recombinant antibody
  * Each vial contains 1mL of study drug
  * The subjects will be treated with A mg/kg once weekly in cohort 2.
  * The Dose A mg/kg will be determined based on the safety, PK, and PD data obtained from previous dose level (cohort 1).
  Interventions: Biological: MG1113
- Cohort 3 (B mg/kg, once weekly) (Active Comparator): * Anti-tissue factor pathway inhibitor (TFPI) recombinant antibody
  * Each vial contains 1mL of study drug
  * The subjects will be treated with B mg/kg once weekly in cohort 3.
  * The Dose B mg/kg will be determined based on the safety, PK, and PD data obtained from previous dose level (cohort 2).
  Interventions: Biological: MG1113

INTERVENTIONS:
Biological: MG1113 — MG1113 subcutaneous (SC) injection

SUMMARY:
The purpose of this study is to assess the safety and tolerability, pharmacokinetics and pharmacodynamics of subcutaneous MG1113 in the multiple ascending dose study in patients with severe hemophilia.

DETAILED DESCRIPTION:
This is a repeat-dose study that assign 5 subjects in each cohort to explore the safety, tolerability, PK, and PD of the study drug by sequentially increasing the study drug.

The route of administration is subcutaneous (SC) injection. Dose escalation will be decided after checking the safety and tolerability at the previous dose to the extent not exceeding the criteria for discontinuation of dose escalation. The dose escalation will be decided by the Steering Committee and Data and Safety Monitoring Boards (DSMB) in the evaluation of the safety and tolerability data obtained from each cohort after repeated administration of MG1113.

The subjects will be treated with 2.0 mg/kg once weekly for 8 weeks in cohort 1. Visit window of ±1 day (calculated from Day1) are allowed for the dosing schedule after first IP administration (Day 1). But next scheduled IP administration must be kept in mind to ensure subjects will not have more than 8 days in between IP dosing interval.

The next dose level (Dose A and B) will be determined based on the safety, PK, and PD data obtained from previous dose level. If a criterion of discontinuation of dose escalation is fulfilled, discussion about dose escalation is available for next cohort. The dose selection and escalation will be finally determined from the Steering Committee and DSMB. The safety, tolerability, PK, and PD data obtained from all subjects up to Cohort 3 will be evaluated by the Steering Committee and Data and Safety Monitoring Boards (DSMB).

ELIGIBILITY:
Inclusion Criteria:

1. Male severe hemophilia A or B patients (FVIII or FIX activity <1%) aged 19-60 years (both inclusive) at screening

   * Patients without inhibitors against FVIII or FIX (having difficulty in their Self-injection of current standard treatment regimen) OR
   * Patients with inhibitors who has a positive inhibitor result of confirmed human factor VIII or IX with an inhibitor titer(≥ 0.6 BU) and failed after ITI treatment or not undergoing ITI
2. ≥50 kg in weight with calculated BMI between 18.5 and 29.9 kg/m^2 (BMI = (Weight [kg])/(height [m])^2)
3. Documentation of ≥4 bleeding episodes (any type or location of bleeds, treated or not) within 6 months prior to screening
4. Agree to use medically acceptable adequate dual contraceptive methods (condom, vasectomy, spermicide, oral contraceptives, intrauterine device, and complete sexual abstinence, etc.) and not to donate sperm until 60 days after administration of the investigational product
5. Voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a detailed explanation on this study and fully understanding the information

Exclusion Criteria:

1. Congenital or acquired anticoagulant disorders other than hemophilia A or B, or conditions of other diseases that increase the risk of bleeding or thrombus (e.g., autoimmune disease)
2. Be at risk of venous thromboembolism or thrombotic microangiopathy per investigator's judgment or have related medical history or family history
3. Be at risk of cardia and/or coronary disease per investigator's judgment or have related medical history or family history
4. Risk factors for venous or arterial disease (e.g., uncontrolled hypertension, uncontrolled diabetes)
5. Any of the following results from laboratory tests:

   * AST(sGOT) or AST(sGPT) > 3 x UNL
   * Total bilirubin > 2 mg/mL
   * Hb < 9.0 g/dL
   * Absolute Neutrophil Count < 1500 /μL
   * Platelet count < 10^5 /μL
   * Have hepatitis B (HBs Ag positive) or C (anti-HCV positive), or have HIV positive test result If the anti-HCV antibody test is positive, the positive hepatitis virus result must be confirmed by a quantitative HCV RNA test
   * Serum Creatinine > 1.5 x Upper limit of normal (ULN)
6. Known or suspected hypersensitivity to the IP or its components
7. Treatment history due to symptoms of fever within 28 days of IP administration or any surgery planned during the study period
8. Clinically significant active chronic disease
9. Subjects who refuse the following wash-out times of Factor VIII, Factor IX, and bypassing agent from the time of first IP administration (Factor VIII: 72 hrs, Factor IX: 96 hrs, Bypassing agent e.g., rFVIIa or aPCC: 96 hrs)
10. Received immune tolerance induction within 30 days prior to administration of the investigational product
11. Received emicizumab within 30 days prior to administration of the investigational product
12. Currently using systemic immunomodulator treatment (e.g., Corticosteroid*, IVIG, interferon or rituximab)

    *High-dose corticosteroids (it is allowed to administer corticosteroid equivalent to up to 20mg/kg daily based on Prednisolone, but if a dose of more is continuously administered in excess of 14 days, it is considered as high dose, such case is excluded from this study. However, inhaled, intranasal, and topical administration of corticosteroids is allowed irrespective of the dose.)
13. Participated in another clinical trial within 30 days of investigational product administration
14. Determined to be ineligible to participate in the study per investigator's judgment due to other reasons including the laboratory test results

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only Male severe hemophilia A or B patients will be enrolled.
Enrollment: 15 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Number of subject with Adverse events, Adverse Drug Reactions, Serious adverse events and Adverse event of special interest (AESI) | Through study completion (Study Day 1 to Day 78 visit)
Incidence of Adverse events, Adverse Drug Reactions, Serious adverse events and Adverse event of special interest (AESI) | Through study completion (Study Day 1 to Day 78 visit)
Severity of Adverse events, Adverse Drug Reactions, Serious adverse events and Adverse event of special interest (AESI) | Through study completion (Study Day 1 to Day 78 visit)
Incidence of injection site reaction | Study Day 1 to Day 57 visit
Severity of injection site reaction | Study Day 1 to Day 57 visit
Number of subjects with abnormal Physical examination | Through study completion (Study Day 1 to Day 78 visit)
Number of subjects with abnormal 12-lead ECG (Ventricular rate in beat/min, Interval for PR in msec, QRS in msec, QTc in msec) | Through study completion (Study Day 1 to Day 78 visit)
Number of subjects with abnormal Vital signs (Blood pressure in mmHg, Pulse rate in beats/min, Respiration rate in breaths/min, Body temperature in ℃) | Through study completion (Study Day 1 to Day 78 visit)
Incidence of clinically significant laboratory value abnormalities | Through study completion (Study Day 1 to Day 78 visit)

SECONDARY OUTCOMES:
Pharmacokinetic assessment - Cmax (Peak plasma concentration) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacokinetic assessment - Cmin (Minimum plasma concentration) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacokinetic assessment - AUC (Area under the plasma concentration versus time curve) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacokinetic assessment - Tmax (Time to maximum plasma concentration after administration) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacokinetic assessment - half-life (T1/2; the time required to reduce the plasma concentration by half) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacokinetic assessment - CL/F (apparent clearance) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacokinetic assessment - Vd/F (apparent volume of distribution) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacokinetic assessment - Accumulation Index (AUCtau_multiple dose/AUCtau_single dose) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Free TFPI in plasma in ng/mL | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Residual TFPI activity in unit/mL | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Diluted PT in sec | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Thrombin generation (Lag time in min) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Thrombin generation (Peak generation in nM) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Thrombin generation (Endogenous thrombin generation potential [ETP] in nM*min) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Pro-coagulant effect (D-dimer in ug/mL) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Pro-coagulant effect (Fibrinogen in mg/dL) | Through study completion (Study Day 1 to Day 78 visit)
Pharmacodynamic assessment - Pro-coagulant effect (Prothrombin fragments 1+2 in pmol/L) | Through study completion (Study Day 1 to Day 78 visit)
Immunogenicity assessment - Any formation of anti-drug antibody (ADA) to MG1113 | Through study completion (Study Day 1 to Day 78 visit)
Efficacy Evaluation - Incidence of new bleeding episode | Study Day 1 to Day 57 visit

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Jin Choi, Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- GC Biopharma Corp., Yongin-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No